CLINICAL TRIAL: NCT06154317
Title: Study for Validation of Target Therapy in Multiple Myeloma Cells From Patients With miRNAs Released From B Cells, and Study of the Bone Marrow Tumor Microenvironment (Microenvironment of MM)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2021-31
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multiple Myeloma (MM) is a hematologic cancer caused by the selective clonal expansion of plasma cells. By acting on the microenvironment of the bone marrow, MM shifts the niche balance and becomes chemoresistant due to its interaction with stromal cells. Despite new therapeutic strategies, MM still remains incurable and new strategies are urgently needed. In order to successfully act on MM, we must use a strategy that reflects its plasticity and blocks it on several targets: proliferation, interaction with the microenvironment, and metastasis.

The main interest of the project is to evaluate the effect of gene therapy identified in vitro, directly on patient-derived samples, in particular to translate the knowledge gained on myeloma cell lines in vitro to primary tumor cells taken from patients.

DETAILED DESCRIPTION:
Multiple Myeloma (MM) is a hematologic cancer caused by the selective clonal expansion of plasma cells. By acting on the microenvironment of the bone marrow, MM shifts the niche balance and becomes chemoresistant due to its interaction with stromal cells. Despite new therapeutic strategies, MM still remains incurable and new strategies are urgently needed. In order to successfully act on MM, we must use a strategy that reflects its plasticity and blocks it on several targets: proliferation, interaction with the microenvironment, and metastasis.

The main interest of the project is to evaluate the effect of gene therapy identified in vitro, directly on patient-derived samples, in particular to translate the knowledge gained on myeloma cell lines in vitro to primary tumor cells taken from patients.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years;
* Diagnosis of multiple myeloma for which a bone marrow biopsy is scheduled for practice
* Patients able to express appropriate consent to participation in the study (e.g., able to understand Italian, patient with intact cognitive abilities).

Exclusion Criteria:

* Absence of signed informed consent form
* Inadequate or insufficient bone marrow biopsy material

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of both sexes with multiple myeloma referred to the SOSD Oncoematologia, Trapianti emopoietici e Terapie cellulari of the CRO in Aviano.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of SOX4 and XBP1 expression in plasma cells from patient with MM | up to 2 years
  Frequencies and 95% confidence interval of SOX4 and XBP1, evaluated in plasma cells from bone biopsies and isolated from bone marrow blood of MM patients by qRT-PCR at different staging.

CONTACTS AND LOCATIONS:
Overall Officials: Mariagrazia Michieli, MD, Principal Investigator — Centro di Riferimento Oncologico (CRO) di Aviano-IRCCS
Locations (1):
- Centro di Riferimento Oncologico (CRO) di Aviano - IRCCS, Aviano, Pordenone, Italy